CLINICAL TRIAL: NCT02429336
Title: Clinical Characteristics of Women Presenting to the Reproductive Endocrinology Clinic
Brief Title: Characteristics of Women With Reproductive Concerns
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01368-XP
Record Dates: First submitted 2015-03-23; First posted 2015-04-29 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Endocrine Disorders of Female Reproductive System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect data that will be generated during an office visit. The data will be gathered and analyzed in research studies that will help with the investigators understanding of various medical conditions.

About 200 subjects will be participating in this study. Participation in this study will not require a patient's time or presence. The medical information contained in a patient's chart from the office visit, including the results of any tests that were ordered at that time, will be transferred to an anonymous database and analyzed together with data from other patients who have similar condition/s.

No follow-up information will be collected. The following information will be collected from a patient's medical record: the medical history and a list of the current medications.

DETAILED DESCRIPTION:
Purpose: To collect the characteristics of patients presenting to the reproductive endocrinology clinic.

Rationale: Patients' characteristics will be analyzed as part of clinical research studies and may help in understanding the causes of their condition.

ELIGIBILITY:
Inclusion Criteria:

* females of childbearing potential experiencing reproductive endocrinology related problems

Exclusion Criteria:

* male or female not of childbearing potential

Min Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population: All patients presenting to the reproductive endocrinology clinic.
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2012-01; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Data collection from patients' charts. | up to 1 year from the time of signing the informed consent for data collection
  Data collection from patients' charts.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Detti, M.D., Principal Investigator — Associate Professor, UTennessee Health Science Center
Locations (1):
- Regional One Health Ob-Gyn Clinic, Memphis, Tennessee, United States